CLINICAL TRIAL: NCT02342509
Title: Automated Control of End-tidal Volatile Anesthetic Concentration Using the MIRUS System: A Comparison of Isoflurane, Sevoflurane and Desflurane in Anesthesia.
Brief Title: Automated Control of End-tidal Volatile Anesthetic Concentration
Acronym: MIRCONTROL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ruhr University of Bochum (Other)
Responsible Party: Principal Investigator, Martin Bellgardt, Dr. med., Ruhr University of Bochum
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: RUB 4780-13
Record Dates: First submitted 2015-01-06; First posted 2015-01-21 (Estimated); Last update posted 2015-01-21 (Estimated); Status verified 2015-01

CONDITIONS: Delayed Recovery From Anesthesia
Keywords: et Control; inhalational sedation; conserve volatile anesthetics
MeSH Terms: conditions — Delayed Emergence from Anesthesia | interventions — Desflurane; Sevoflurane; Isoflurane

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Desflurane (Experimental): Desflurane 5.0-6.0 Vol% (1.0 MAC) in Oxygen (FiO2 0.8-0.95)
  Interventions: Drug: Desflurane
- Sevoflurane (Experimental): Sevoflurane 1.4-2.1 Vol% (1.0 MAC) in Oxygen (FiO2 0.8-0.95)
  Interventions: Drug: Sevoflurane
- Isoflurane (Active Comparator): Isoflurane 0.9-1.2 Vol% (1.0 MAC) in Oxygen (FiO2 0.8-0.95)
  Interventions: Drug: Isoflurane

INTERVENTIONS:
Drug: Desflurane — Group A: Desflurane 5.0-6.0 Vol% (1.0 MAC) in Oxygen (FiO2 0.8-0.95)
  Other Names: Suprane
  Arms: Desflurane
Drug: Sevoflurane — Group B: Sevoflurane 1.4-2.1 Vol% (1.0 MAC) in Oxygen (FiO2 0.8-0.95)
  Other Names: Sevorane
  Arms: Sevoflurane
Drug: Isoflurane — Group C: Isoflurane 0.9-1.2 Vol% (1.0 MAC) in Oxygen (FiO2 0.8-0.95)
  Other Names: Forene
  Arms: Isoflurane

SUMMARY:
The new MIRUS system as well as the established AnaConDa system uses a reflector to conserve volatile anaesthetics (VA). Both systems act with commercially available ICU ventilators. In contrast to AnaConDa the MIRUS includes an automated control of end-tidal VA concentrations. In this study the investigators compared feasibility, costs and recovery times after anaesthesia with isoflurane (ISO), sevoflurane (SEVO) or desflurane (DES) in ventilated and spontaneously breathing patients.

DETAILED DESCRIPTION:
The study was approved by the appropriate Institutional Review Board. After written informed consent 63 ASA I-III patients undergoing elective hip or knee replacement surgery under general anesthesia were included. Patients were randomly organized into 3 groups (20-22 each). Anesthesia was induced with intravenous anaesthetics. After tracheal intubation MIRUS automatically adjusted the end-tidal VA concentration to 1.0 MAC. Patients were ventilated with the Puritan Bennett 840 ICU ventilator. After 1 h of anaesthesia with 1.0 MAC the ventilator mode was switched from SIMV V+ (totally controlled ventilation, "passive patient", with a tidal volume of 8 ml/IBW) to proportional assist ventilation (PAV) with 50% support ("active patient"). At the end of surgery the MIRUS system was stopped (MAC set to 0.0) and recovery times were measured.

ELIGIBILITY:
Inclusion Criteria:

* Signing of the informed consent document (patient or relatives).
* Patient age 18 years or older.
* ASA I-III

Exclusion Criteria:

* ASA IV patients
* Epidural or spinal analgesia
* Allergy or known hypersensitivity to any of the study drugs
* Patients with known or suspected genetic susceptibility to malignant hyperthermia
* Previous participation in this trial
* Participation in another clinical trial within 4 weeks prior to selection.
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2014-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
volatile anaesthetics (VA) consumption | duration of anesthesia: max. 3 h

SECONDARY OUTCOMES:
recovery times | duration post anesthesia care: max. 8 h after anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Weber, PhD, Principal Investigator — Ruhr-Universtiy of Bochum, Germany

REFERENCES:
- [Background] Bomberg H, Glas M, Groesdonk VH, Bellgardt M, Schwarz J, Volk T, Meiser A. A novel device for target controlled administration and reflection of desflurane--the Mirus. Anaesthesia. 2014 Nov;69(11):1241-50. doi: 10.1111/anae.12798. Epub 2014 Jul 9. PMID 25040673
- [Background] Meiser A, Sirtl C, Bellgardt M, Lohmann S, Garthoff A, Kaiser J, Hugler P, Laubenthal HJ. Desflurane compared with propofol for postoperative sedation in the intensive care unit. Br J Anaesth. 2003 Mar;90(3):273-80. doi: 10.1093/bja/aeg059. PMID 12594136